CLINICAL TRIAL: NCT03334019
Title: Prevalence and Risk Factors for Coxiella Burnetii Seropositivity (Q Fever) Among Adults in Western France
Acronym: MEDVETFQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: ONIRIS (Industry)
Responsible Party: Sponsor
Other Study IDs: RC16_0420
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Q Fever
MeSH Terms: conditions — Q Fever | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the participants in the study will provide a blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects: Data collected on general population, farmers and veterinarians though questionnaires and blood samples.
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test — Data collected on general population, farmers and veterinarians though questionnaires and blood samples.

SUMMARY:
Diseases naturally transmitted between animals and humans (zoonoses) are one of the leading causes of emergence or re-emergence of human infectious diseases. Non-foodborne zoonoses are commonly transmitted to human directly by contact with infected animals or contaminated environment. People working with animals such as farmers and veterinarians are particularly at risk of infection. Some zoonoses can also be transmitted indirectly thought the air and therefore can affect the general population. Example is Q fever, a disease caused by Coxiella burnetii, a bacterium highly resistant in the environment.

In Western France, Q fever is endemic in cattle herds. To improve human zoonotic disease surveillance, the investigators will conduct a population based study in this area.

The aims of the study are:

1. To assess seroprevalence of Coxiella burnetii infection among general population, farmers and veterinarians in Western France
2. To identify risk factors for Coxiella burnetii seropositivity in these populations

DETAILED DESCRIPTION:
In order to estimate seroprevalence and risk factors for Coxiella burnetii infection in humans, the investigators will conduct a cross-sectional study in three groups:

* blood donors at blood donation organizations (general population)
* beef and dairy cattle farmers
* veterinarians involved in a rural practice

All the participants in the study will provide a blood sample and will fill in a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Give a written informed consent
* Be 18 years old and over
* Be able to speak French

Exclusion Criteria:

* Adults under protection (guardianship or curators)
* Contraindication for drawing blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * blood donors at blood donation organizations (general population)
  * beef and dairy cattle farmers
  * veterinarians involved in a rural practice
Sampling Method: Non-Probability Sample
Enrollment: 559 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Antibody titers against Coxiella burnetii in general population in Western France | Day 0
  Blood samples will be taken on blood donors for detection of Coxiella burnetii antibodies by indirect immunofluorescence assay.
Antibody titers against Coxiella burnetii in farmers population in Western France | Day 0
  Blood samples will be taken on farmers for detection of Coxiella burnetii antibodies by indirect immunofluorescence assay.
Antibody titers against Coxiella burnetii in veterinarians population in Western France | Day 0
  Blood samples will be taken on veterinarians for detection of Coxiella burnetii antibodies by indirect immunofluorescence assay.

SECONDARY OUTCOMES:
Measure of association between Coxiella burnetii seropositivity risk and socio-demographic | Day 0
  A short questionnaire will be filled in by participants (general population) to collect socio-demographic, lifestyle and occupational factors.
Measure of association between Coxiella burnetii seropositivity risk and lifestyle | Day 0
  A short questionnaire will be filled in by participants (farmers) to collect socio-demographic, lifestyle and occupational factors.
Measure of association between Coxiella burnetii seropositivity risk and occupational factors. | Day 0
  A short questionnaire will be filled in by participants (veterinarians) to collect socio-demographic, lifestyle and occupational factors.
Measure of association between Coxiella burnetii seropositivity in humans (general population) and cattle herds' prevalence of Coxiella burnetii infection. | Day 0
  Besides blood samples taken on participants, blood samples and milk samples will be taken on beef and dairy cattle herds, respectively, to determine the prevalence of Coxiella burnetii infection in cattle herds.
Measure of association between Coxiella burnetii seropositivity in humans (farmers) and cattle herds' prevalence of Coxiella burnetii infection. | Day 0
  Besides blood samples taken on participants, blood samples and milk samples will be taken on beef and dairy cattle herds, respectively, to determine the prevalence of Coxiella burnetii infection in cattle herds.
Measure of association between Coxiella burnetii seropositivity in humans ( veterinarians) and cattle herds' prevalence of Coxiella burnetii infection. | Day 0
  Besides blood samples taken on participants, blood samples and milk samples will be taken on beef and dairy cattle herds, respectively, to determine the prevalence of Coxiella burnetii infection in cattle herds.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Moret, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France